CLINICAL TRIAL: NCT02795416
Title: A 16-week, Single Arm, Multicenter Study for the Assessment of Efficacy and Safety of Secukinumab in aduLt Patients With Moderate to Severe plaquE Psoriasis in Turkish Population
Brief Title: Assessment of Efficacy and Safety of Secukinumab in Adult Patients in Turkish Population
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457ATR01
Record Dates: First submitted 2016-05-16; First posted 2016-06-10 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Psoriasis
Keywords: Moderate to severe plaque psoriasis, PASI, secukinumab, monoclonal antibody, Turkish population
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- "Secukinumab" "Cosentyx TM" (Experimental): "Secukinumab" "Cosentyx TM" 150 mg PFS (pre-filled syringe) containing for solution for s.c. injection will be applied as 2 units (300 mg dosage) per patient at each visit.
  First month: 300 mg injections/week, 4 weeks Starting from 4th week until Week 16, one injection/month
  Interventions: Drug: "Secukinumab" "Cosentyx TM"

INTERVENTIONS:
Drug: "Secukinumab" "Cosentyx TM" — "Secukinumab" "Cosentyx TM" 150 mg PFS (pre-filled syringe) containing for solution for s.c. injection will be applied as 2 units (300 mg dosage) per patient at each visit.
  First month: 300 mg injections/week, 4 weeks Starting from 4th week until Week 16, one injection/month

SUMMARY:
Secukinumab targets a different interleukin and has potential to be used as alternative to existing treatments. This study will provide clinical data with respect to efficacy through Psoriasis Area and Severity Index (PASI) at 16 weeks, safety/tolerability of secukinumab and evaluate the impact of the treatment on quality of life and work productivity in subjects with moderate to severe plaque psoriasis in the Turkish population.

DETAILED DESCRIPTION:
To demonstrate the efficacy of secukinumab in subjects with moderate to severe plaque psoriasis based on the percentage of PASI 90 responder patients at Week 16 as compared to baseline Evaluation of onset of efficacy measured by the percentage of patient achieving PASI 75 and PASI 90 at week 4 The efficacy of treatment using Investigator's Global Assessment modified 2011 (IGA mod 2011) at week 4 and week 16 Work productivity (measured with WPAI-PSO) at Week 16 Changes in quality of life measured with the Dermatology Life Quality Index (DLQI) at Week 16 Health assessment questionnaire -Disability index (HAQ-DI) in patients with psoriatic arthritis (PsA)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand and comply with the requirements of the study and communicate with the investigator
* Diagnosis of chronic plaque psoriasis for at least 6 months before enrollment
* Patients who were evaluated as candidates for systemic therapy, defined as having psoriasis intolerant or /and inadequately controlled by: topical treatment (including topical corticosteroid) and/or phototherapy and/or any previous systemic treatment for psoriasis or any previous treatment with biologic agents

Exclusion Criteria:

* Forms of psoriasis other than plaque psoriasis
* Drug-induced psoriasis
* Previous exposure to secukinumab or any other biologic drug directly targeting IL-17A or IL-17RA
* Pregnant or nursing (lactating) women
* Active ongoing inflammatory diseases other than psoriasis or psoriatic arthritis that might confound the evaluation of the benefit of secukinumab
* Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions)
* Pre-existing or recent-onset central or peripheral nervous system demyelinating disorders
* Significant medical problems, including but not limited to the following: uncontrolled hypertension, congestive heart failure
* Active systemic infections during the 2 weeks prior to enrollment
* History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection
* Past medical history record of, or current infection with, human immunodeficiency virus (HIV), hepatitis B or hepatitis C prior to enrollment
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years
* History or evidence of ongoing alcohol or drug abuse, within the last 6 months prior to enrollment
* Plans for administration of live vaccines during the study period or in the 6 weeks prior to enrollment
* Not willing to limit UV light exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of PASI 90 responder patients at Week 16 as compared to baseline | 16 week
  The primary endpoint has been chosen as percentage of PASI 90 responder patients. PASI 90 is accepted as clear or almost clear of psoriatic lesions which are the ultimate goal of treatment in plaque psoriasis.

SECONDARY OUTCOMES:
Evaluation of onset of efficacy measured by the percentage of patient achieving PASI 75 and PASI 90 at week 4 | 4 week
  Patients, who achieved PASI 75 and PASI 90 response at week 4 will be counted by using frequencies and percentages (a subject is defined as a PASI 90 responder if the PASI score is reduced by 90% or more compared to baseline visit)
The efficacy of treatment using Investigator's Global Assessment modified 2011 (IGA mod 2011) at week 4 and week 16 | 4 and 16 week
  Investigator's Global Assessment (IGA mod 2011) score will be explained by using descriptive statistics at week 4 and week 16. Change between week 4 and week 16 comparing to baseline
Work productivity (measured with WPAI-PSO) at Week 16 | 16 week
  Work productivity (WPAI-PSO) at week 16 will be evaluated by using descriptive statistics at week 16. Changes at work productivity through the visits will be inspected by using Repeated Measures ANOVA test.
Changes in quality of life measured with the Dermatology Life Quality Index (DLQI) at Week 16 | 16 week
  Changes in quality of life measured with Dermatology Life Quality Index (DLQI) through visits will be evaluated by using Repeated Measures ANOVA test.
Health assessment questionnaire -Disability index (HAQ-DI) in patients with psoriatic arthritis (PsA) | 16 week
  Health Assessment Questionnaire-Disability Index (HAQ-DI) will be evaluated at all visits by using descriptive statistics. The change between visits will be evaluated by Repeated Measures ANOVA test.

OTHER OUTCOMES:
In case of insulin resistance determined at the baseline, the change in the resistance level as measured by HOMA-IR | 16 week
  Change in HOMA-IR level between baseline and week 16 will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Atakan, Prof.Dr, Study Director — Hacettepe University Medical Faculty; Server Serdaroglu, Prof.Dr, Study Director — Istanbul University Cerrahpasa Medical Faculty; Emel Bulbul Baskan, Prof.Dr, Principal Investigator — Uludag University Medical Faculty; Erkan Alpsoy, Prof.Dr, Principal Investigator — Akdeniz University Medical Faculty; Ferda Artuz, Prof.Dr, Principal Investigator — Ankara City Hospital Bilkent; Guliz Ikizoglu, Prof.Dr, Principal Investigator — Mersin University Medical Faculty; Guzin Ozarmagan, Prof.Dr, Principal Investigator — Istanbul University Istanbul Medical Faculty; Ilgen Ertam, Prof.Dr, Principal Investigator — Ege University Medical Faculty; Murat Borlu, Prof.Dr, Principal Investigator — Erciyes University Medical Faculty; Muzeyyen Sanlı Gonul, Ass.Prof, Principal Investigator — Dıskapi Training and Research Hospital; Nilgun Senturk, Prof.Dr, Principal Investigator — Ondokuz Mayıs University Medical Faculty; Savas Yaylı, Ass.Prof, Principal Investigator — Karadeniz Technical University; Serhat Inaloz, Prof.Dr., Principal Investigator — Gaziantep University Medical Faculty; Sinan Dogan, Spec.Dr, Principal Investigator — Bozyaka Training and Research Hospital; Tulin Ergun, Prof.Dr, Principal Investigator — Marmara university Medical Faculty